CLINICAL TRIAL: NCT05648838
Title: The Study for Evaluation of Safety and Efficacy of Pivot Balloon to Monitoring Acute RV Failure and Reduction of Functional Tricuspid Regurgitation : Multi-center, Open Label, Single Arm, Investigator Initiated Exploratory Pilot Study
Brief Title: Evaluation of Safety and Efficacy of Pivot Balloon to Monitoring Acute RV Failure and Reduction of FTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Seung-Whan Lee,MD,PhD, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pivot Balloon-FIM
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Functional Tricuspid Regurgitation
Keywords: FTR; RV failure; TauPnu

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pivot Balloon (Experimental): mornitoring with transcatheter Tricuspid Regurgitation reduction system
  Interventions: Device: Pivot Balloon Catheter

INTERVENTIONS:
Device: Pivot Balloon Catheter — mornitoring acute RV failure and reduction of Functional Tricuspid Regurgitation

SUMMARY:
Pivot Balloon to monitoring acute RV failure and reduction of Functional Tricuspid Regurgitation

DETAILED DESCRIPTION:
The study for evaluation of safety and efficacy of Pivot Balloon to monitoring acute RV failure and reduction of Functional Tricuspid Regurgitation : multi-center, open label, single arm, investigator initiated exploratory pilot study

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 20 years or above
* Target of Thoracic Surgery for TR and patients above the severe level on the criteria presented in the Classification of TR Grade based on echocardiogram, among those with TR, for whom a surgical treatment has been decided
* An individual who voluntarily agreed to the participation in the clinical trial and signed the written consent
* An individual who is able to understand and comply with the instructions and who can participate in the period before the clinical trial

Exclusion Criteria:

* Uncontrolled hyperthyroidism
* A recent formation of soft blood clot or embolic material
* Uncorrected coagulopathy
* Prohibition of anticoagulant agents
* Previous insertion of a device such as an Implantable Cardioverter Defibrillator (ICD) or a pacemaker
* Presence of malignant tumor or benign tumor such as myxoma in the heart
* Presence of a symptom of active infection
* Chronic pulmonary disease
* Congenital tricuspid valve insufficiency
* Pregnant or lactating mother, or a female patient planning pregnancy during the period of clinical trial, or a female not using an approved contraceptive with the possibility of pregnancy
* Participation in another clinical trial 30 days prior to the screening
* In addition, anyone showing a clinical finding deemed to be unsuitable for the clinical trial by the Principal Investigator or the Investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
change of tricuspid regurgitation grade (1) | immediately after the procedure
  check the success of surgery /measure the size of the TR area
change of tricuspid regurgitation grade (2) | immediately after the procedure
  examine the changes in the severity of tricuspid valve insufficiency with Echocardiogram

SECONDARY OUTCOMES:
change of tricuspid regurgitation valve hemodynamics | within 24 h of insertion
  examine the changes in the severity of tricuspid valve insufficiency with Echocardiogram
evaluate the efficacy based on the function of early diagnosis (1) | within 24 h of insertion
  examine tricuspid regurgitation intolerance
evaluate the efficacy based on the function of early diagnosis (2) | within 24 h of insertion
  evaluate the technical success rate of the implantation and the technical feasibility of 'Pivot Balloon'

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Whan Lee, PhD, Principal Investigator — Asan Medical Center
Locations (10):
- South Korea (10):
  - Keimyung University Dongsan Hospital, Daegu, Dalseo-gu
  - Hallym University Medical Center, Anyang, Dongan-gu
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Chungnam National University Hospital (CNU Hospital), Daejeon, Jung-gu
  - Yeungnam University Hospital, Daegu, Nam-gu
  - Ulsan Hospital, Ulsan, Nam-gu
  - Chungnam National University Sejong Hospital, Sejong, Sejong-si
  - Asan Medical Center, Seoul, Songpa-gu
  - Bucheon Sejong Hospital, Bucheon-si
  - Samsung Medical Center, Seoul

REFERENCES:
- [Background] Downie IP, Evans BT. Re: Holmes S, Hutchison I. Reconstruction of the orbital floor after its removal for malignancy. Br J Oral Maxillofac Surg 2001; 39: 158-159. Br J Oral Maxillofac Surg. 2001 Dec;39(6):485. doi: 10.1054/bjom.2001.0679. No abstract available. PMID 11735152
- [Derived] Kim EK, Chon MK, Kim HS, Park YH, Lee SH, Choo KS, Je HG, Kim DH, Kim TO, Koh YS, Park JH, Lee JH, Choi YJ, Shin ES, Yoon HJ, Lee SW, Hahn JY. Safety and Efficacy of Pivot-Balloon for Severe Tricuspid Regurgitation: The First-in-Man Experiences. Korean Circ J. 2025 Jan;55(1):20-31. doi: 10.4070/kcj.2024.0147. Epub 2024 Oct 14. PMID 39601393